CLINICAL TRIAL: NCT01398813
Title: Survey of X-Linked Hypohidrotic Ectodermal Dysplasia Carrier Women's Outlook Towards Reproduction, Potential XLHED Treatments and Genetic Testing
Brief Title: X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED) Carrier Outlook Toward Reproduction Survey
Acronym: X-CORS
Status: Completed | Type: Observational
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ECP-008
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Hypohidrotic Ectodermal Dysplasia; X-Linked Hypohidrotic Ectodermal Dysplasia
Keywords: HED; XLHED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
In this survey of X-Lined Hypohidrotic Ectodermal Dysplasia (XLHED) carrier females, Edimer proposes to review responses to an XLHED Carrier Outlook toward Reproduction Survey in order to understand attitudes toward reproduction, potential treatments and genetic testing in order to improve the understanding of the decisions that XLHED carrier females make regarding their reproductive future.

DETAILED DESCRIPTION:
The full survey is available here: https://www.surveymonkey.com/s/X-CORS

For more questions or more details you may contact the Principal Investigator, Carrie Milliard: MILLIC@mmc.org or 207-662-6712

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent;
2. 18 years of age or older
3. Females with:

   * the clinical characteristics of HED, including at least two of the following characteristics:

     * clinical signs and symptoms of HED:

       * a history of decreased sweating;
       * abnormal teeth (fewer permanent teeth, teeth are smaller than average and often have conical crowns);
       * sparseness of scalp and body hair;
   * AND

     * a clinical diagnosis from a healthcare professional;
     * or at least one HED affected family member
   * OR genetically confirmed HED or XLHED;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll XLHED carrier females
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To study the outlook of XLHED carrier females toward reproduction, potential XLHED treatments and genetic testing. | study day 1
  Survey results will be collected during the 1 day of subject involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Milliard, CGC, Principal Investigator — Maine Medical Partners Pediatric Specialty Care
Locations (1):
- Carrie Milliard, Portland, Maine, United States